CLINICAL TRIAL: NCT04663789
Title: Efficacy of Routine Staple Line Reinforcement Versus no Reinforcement on Pancreatic Fistula After Minimally Invasive Distal Pancreatectomy: A Single Center, Parallel, Randomized Controlled Trial
Brief Title: Routine Staple Line Reinforcement for Minimally Invasive Distal Pancreatectomy
Acronym: Double-Lock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Feng Tian, Attending, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PUMCHTF2
Record Dates: First submitted 2020-11-24; First posted 2020-12-11 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Pancreas Neoplasm; Stump; Surgery--Complications
Keywords: Staple line; Reinforcement; Pancreatic fistula
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Intervention Model Description: The study is a single-center, randomized controlled clinical trial. Grouping: the study group is set as "staple line plus reinforcement" group, in which a lock stitch will be placed after transecting the pancreas with stapler. While the control group is set as "staple line with no reinforcement" group, in which no additional reinforcement is used after transecting the pancreas with stapler.
Who Masked: Participant, Outcomes Assessor
Masking Description: It will be single blinded. Operator, first assistant and data collector could not be blinded. Whereas patients, nurses, data analyzer, and those who have the access to the primary predictor will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staple line plus reinforcement (Experimental): In this experimental group, a lock stitch will be placed after transecting the pancreas with stapler.
  Interventions: Procedure: reinforcement of the staple line
- staple line with no reinforcement (Other): In this control group, no additional reinforcement is used after transecting the pancreas with stapler.
  Interventions: Procedure: staple only

INTERVENTIONS:
Procedure: reinforcement of the staple line — The operator will perform reinforcement of the staple line with a continuous lock stitch.
  Arms: Staple line plus reinforcement
Procedure: staple only — The operator transect the pancreas with stapler only, without staple line reinforcement.
  Arms: staple line with no reinforcement

SUMMARY:
Postoperative fistula is the major complications of distal pancreatectomies which prohibit patients' recovery. Previous studies have reported controversial results regarding the efficacy of pancreatic stump reinforcement methods. Prior research has commonly included minimally invasive and open cases together. Moreover, stapler and suture were combined in most studies making interpretation difficult. Data has shown that staple line plus reinforcement might potentially decrease the CR-POPF rate of patients who underwent distal pancreatectomies, but well-designed high-quality evidence is lacking. Thus, the investigators design the present study to the question that whether routine staple line plus reinforcement would bring benefit for participants.

DETAILED DESCRIPTION:
Distal pancreatectomy (DP)is the standard surgical method for benign or malignant pancreatic tumors locating at body and tail [1]. Clinically relevant postoperative pancreatic fistula (CR-POPF) is the major complication after pancreatectomy. In literature, reported CR-POPF rate after distal pancreatectomy varied between 5% and 64% from different centers. It's still a challenge to prevent CR-POPF via effective pancreatic remnant closure and no consensus on the optimal surgical technique has been established. Reported surgical strategies to prevent CR-POPF included stapler transection, staple line reinforcement, stump coverage with autologous tissue or fibrin glue, mesh reinforcement, and prophylactic administration of octreotide. However, none had convincing outcome [2-4].

Data has shown that staple line plus suture reinforcement might potentially decrease the CR-POPF rate of patients who underwent distal pancreatectomies, but well-designed high-quality evidence is lacking. Meanwhile, prior researches have commonly included minimally invasive and open cases together. Moreover, stapler and suture were combined in most studies making interpretation difficult [5-8].

Thus, the investigators design a single-centered, parallel, randomized controlled trial to compare the efficacy of routine staple line plus reinforcement versus staple only on the CR-POPF rate of participants who underwent minimally invasive distal pancreatectomies.

ELIGIBILITY:
Inclusion Criteria:

* Those who will receive distal pancreatectomy via minimally invasive approaches, no matter benign or malignant;
* Aged from 18 - 80 years;
* Preoperative diagnosis of serous or mucinous cystic adenoma;
* Preoperative diagnosis of solid pseudopapillary tumor (SPT);
* Preoperative diagnosis of neuroendocrine tumor;
* Preoperative diagnosis of intraductal papillary mucinous neoplasm (IPMN);
* Preoperative diagnosis of or pseudocyst;
* Preoperative diagnosis of distal pancreatic malignancies;
* Patients willing to provide informed consent.

Exclusion Criteria:

* History of upper abdominal surgical history such as splenectomy, gastrectomy, liver resection, duodenal or pancreatic resection (not including laparoscopic cystectomy);
* Pancreatic trauma;
* With pneumoperitoneum contraindications;
* With severe heart or pulmonary diseases which is not fit for surgeries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant postoperative pancreatic fistula (CR-POPF) | Postoperative postoperative day 30.
  CR-POPF is defined according to the revised 2016 version of ISGPS (International Study Group on Pancreatic Surgery) classification and grading of POPF. A CR-POPF is defined as a drain output of any measurable volume of fluid with amylase level greater than 3 times the upper Institutional normal serum amylase level, associated with a clinically relevant development/condition related directly to the POPF.

SECONDARY OUTCOMES:
Operative time | Postoperative postoperative day 30.
  Skin-to-skin time
Estimated blood loss | Postoperative postoperative day 30.
  Total blood loss during surgery
Length of postoperative hospital stay | Postoperative postoperative day 30.
  Days of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Guo, Doctor, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China